CLINICAL TRIAL: NCT01357044
Title: An Extract of Pomegranate Fruit and Galangal Rhizome Increases the Numbers of Motile Sperm: A Prospective, Randomised, Controlled, Double-Blinded Trial
Brief Title: Effects of Plant Extracts on Semen Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horsens Hospital (Other)
Collaborators: Videns- og Forskningscenter for Alternativ Behandling (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, Horsens Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LRB-SU-010
Record Dates: First submitted 2011-05-17; First posted 2011-05-20 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Poor Semen Quality
Keywords: Semen quality; Plant extracts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plant extracts (Active Comparator)
  Interventions: Dietary Supplement: Extracts of Punica granatum and Alpinia galanga
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Extracts of Punica granatum and Alpinia galanga — Tablets, two in the morning and two in the evening
  Arms: Plant extracts
Dietary Supplement: Placebo — Tablets, two in the morning and two in the evening
  Arms: Placebo

SUMMARY:
this is a prospective randomized placebo-controlled double-blinded trial investigating the effect of plant extracts from Alpinia galanga and Punica granatum on human semen quality. The investigators hypothesize that these plant extracts will improve semen quality.

ELIGIBILITY:
Inclusion Criteria:

* Reduced semen quality

Exclusion Criteria:

* Total count of motile sperm less than 1 million sperm/ejaculate or more than 200 million sperm/ejaculate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Count of motile sperm per ejaculate | Each participant is given plant extract for three months with flanking semen analyses.

SECONDARY OUTCOMES:
Morphology: percentage of morphologically abnormal sperm in the ejaculate | Each participant is given plant extract for three months with flanking semen analyses.
  If we find an increase in the primary outcome measure in data from participants receiving plant extracts and not in those receiving placebo tablets, we wish to further investigate whether sperm morphology also improves when consuming the plant extracts, e.g. whether the percentage of abnormal sperm in an ejaculate decreases in the group of participants receiving the active plant extracts

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Reproductive Biology, Horsens, Denmark

REFERENCES:
- [Derived] Fedder MD, Jakobsen HB, Giversen I, Christensen LP, Parner ET, Fedder J. An extract of pomegranate fruit and galangal rhizome increases the numbers of motile sperm: a prospective, randomised, controlled, double-blinded trial. PLoS One. 2014 Oct 2;9(9):e108532. doi: 10.1371/journal.pone.0108532. eCollection 2014. PMID 25275520